CLINICAL TRIAL: NCT07220603
Title: An Open-Label Extension Study Evaluating Safety and Pharmacokinetics in Participants With Myotonic Dystrophy Type 1 (FREEDOM-OLE)
Brief Title: An Open-Label Extension Study of PGN-EDODM1 in People With Myotonic Dystrophy Type 1 (FREEDOM-OLE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PepGen Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGN-EDODM1-103
Record Dates: First submitted 2025-10-22; First posted 2025-10-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Myotonic Dystrophy 1
Keywords: DM1; Myotonic Dystrophy 1; Myotonic Dystrophy; PepGen; PGN-EDODM1; Myotonic Muscular Dystrophy; Steinhert's Disease; Myotonic Dystrophies; Genetic Diseases, Inborn; Neuromuscular Diseases; Nervous System Diseases; Musculoskeletal Diseases; Myotonic Disorders; Muscular Disorders, Atrophic; Heredodegenerative Disorders, Nervous System; Muscular Diseases
MeSH Terms: conditions — Myotonic Dystrophy; Genetic Diseases, Inborn; Neuromuscular Diseases; Nervous System Diseases; Musculoskeletal Diseases; Myotonic Disorders; Muscular Disorders, Atrophic; Heredodegenerative Disorders, Nervous System; Muscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PGN-EDODM1 (Experimental): Participants will receive doses of PGN-EDODM1 once every 4 weeks (Q4W)
  Interventions: Drug: PGN-EDODM1

INTERVENTIONS:
Drug: PGN-EDODM1 — Administered by intravenous (IV) infusion

SUMMARY:
The purpose of this study is to learn about the long-term safety and tolerability of PGN-EDODM1 in participants with myotonic dystrophy type 1 (DM1) who have completed a prior study with PGN-EDODM1.

ELIGIBILITY:
Inclusion Criteria:

* Participant has completed a prior study with PGN-EDODM1

Exclusion Criteria:

* Abnormal laboratory tests at screening considered clinically significant by the Investigator
* Use of an investigational drug (other than PGN-EDODM1), device, or product, within 30 days or 5 half-lives of the study drug (whichever is longer) prior to study entry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by number of participants with Adverse Events (AEs) | Baseline through Week 108

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - CIUSSS du Saguenay-Lac-Saint-Jean, Saguenay